CLINICAL TRIAL: NCT07312305
Title: Small Airways Disease Functional Assessment in Idiopathic Pulmonary Fibrosis (SWIFT-IPF)
Acronym: SWIFT-IPF
Status: Recruiting | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Michele Mondoni, MD, Associated Professor of Respiratory Medicine, University of Milan
Other Study IDs: SWIFT-IPF
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Pulmonary Fibrosis; Small Airways Disease
Keywords: IPF; SAD; SBW-N₂
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IPF: IPF of any severity degree, diagnosed according to the 2022 ATS/ERS/JRS/ALAT guidelines

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a chronic, fibrosing, and progressive lung disease of unknown cause, whose incidence increases proportionally from the age of 60. It is characterized by a poor prognosis. Antifibrotic therapy can slow the progression of the disease and reduce mortality, but the life expectancy is less than 7-10 years in the vast majority of patients with IPF. There are no studies in the literature that have evaluated the presence of small airway disease in patients with IPF prior to the initiation of pharmacological therapy, using the nitrogen washout test. This test is currently considered the only non-invasive method capable of detecting ventilation inhomogeneity and closing volume, which are indicators of small airway dysfunction. The investigators carried out an Italian prospective, observational, multicenter study with the primary aim to assess the prevalence of small airway disease measured by the nitrogen washout test (evaluating the following functional parameters: phase 3 slope, closing volume, closing capacity, closing volume/vital capacity, closing capacity/total lung capacity, and phase 4 slope) in a group of patients with IPF at the time of diagnosis, before the initiation of antifibrotic therapy. During outpatients visits clinical, functional and radiological data will be collected. Results will be compared to an healthy control group matched with IPF population. Variations in small airways disease parameters will be assessed after one year of antifibrotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* IPF of any degree of severity, diagnosed according to the 2022 ATS/ERS/JRS/ALAT guidelines

Exclusion Criteria:

* Refusal to participate in the study
* Patients unable to provide informed consent for participation in the study
* IPF exacerbation in the 6 months prior to enrollment
* Previous diagnosis of chronic airway disease (e.g., bronchial asthma, chronic obstructive bronchitis, bronchiectasis with a cause other than IPF)
* Presence of bronchial obstruction defined by an FEV1/FVC (or FEV1/VC) ratio below the lower limit of normal
* Chronic therapy with long-acting bronchodilators or combinations of bronchodilators and inhaled corticosteroids
* Inability of the patient to perform reproducible pulmonary function tests
* Chronic treatment with systemic corticosteroids or immunosuppressants
* Concomitant lung or pleural cancer
* Pregnancy or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPF of any severity diagnosed according to the 2022 ATS/ERS/JRS/ALAT guidelines, attending the specialist outpatient clinics of the Pulmonology Units of ASST Santi Paolo e Carlo and ASST Fatebenefratelli-Sacco (Milan, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of small airway disease in a group of patients with IPF at the time of diagnosis, before the initiation of antifibrotic therapy. | 1 year
  To evaluate the percentage of patients with IPF at the time of diagnosis, before the initiation of antifibrotic therapy, with small airway disease measured by the nitrogen washout test (assessing the following functional parameters: phase 3 slope, closing volume, closing capacity, closing volume/vital capacity, closing capacity/total lung capacity, and phase 4 slope).

SECONDARY OUTCOMES:
Relationship between computed tomography (CT) features and functional parameters indicative of small airway disease. | 1 year
  To evaluate the relationship between CT features (radiologic pattern type, presence/absence of mediastinal lymphadenopathy, presence/absence of any type of emphysema involving ≥5% of total lung volume, extent of disease, disease progression, air trapping, black lung) and functional parameters indicative of small airway disease.
To compare the indices of small airway dysfunction and the prevalence of small airway disease in patients with IPF and age-matched healthy subjects | 1 year
  To compare the indices of small airway dysfunction and the prevalence of small airway disease in patients with IPF and age-matched healthy subjects (without respiratory comorbidities).
Relationship between clinical and epidemiological characteristics of the cohort and the presence and severity of small airway disease | 1 year
  To study the relationship between clinical and epidemiological characteristics of the cohort and the presence and severity of small airway disease
Prevalence of small airway disease in patients with IPF and concomitant emphysema with patients with IPF alone | 1 year
  To compare the prevalence of small airway disease in patients with IPF and concomitant emphysema (combined pulmonary fibrosis and emphysema, CPFE), defined as the presence of any type of emphysema involving ≥5% of total lung volume, with patients with IPF alone.
Correlation between functional characteristics, parameters of small airway dysfunction and fibrosis extent indices on chest CT-scan | 1 year
  To evaluate the correlation between functional characteristics: forced expiratory flow at 25-75% of vital capacity (FEF25-75), forced vital capacity (FVC) and diffusing of the lung for carbon monoxide (DLCO) with parameters of small airway dysfunction from the Single Breath Nitrogen (SBN2) test, as well as disease extent indices on chest CT-scan
Relationship between exercise performance and the presence and severity of small airway disease | 1 year
  To evaluate the relationship between exercise performance (meters, oxygen saturation nadir), assessed by the six-minute walk test distance, and the presence and severity of small airway disease
Relationship between dyspnea degree and the presence and severity of small airway disease. | 1 year
  To evaluate the relationship between the degree of dyspnea, measured by the modified Medical Research Council (mMRC) scale, and the presence and severity of small airway disease.
Clinical and functional characteristics of IPF patients with different alterations in the DLCO subcomponents | 1 year
  To evaluate the clinical and functional characteristics of IPF patients with different alterations in the DLCO subcomponents (alveolar volume - VA <80% predicted, Transfer Coefficient of CO - KCO <80% predicted, ventilation inhomogeneity - VA/Total Lung Capacity (TLC) <0.8)
Relationship between different scores as the GAP index, CPI, KBILD and UCSD Shortness of Breath Questionnaire, and the presence and severity of small airway disease | 1 year
  To evaluate the relationship between different scores as the Gender Age Physiology (GAP) index, Composite Physiologic Index (CPI) , the King's Brief Interstitial Lung Disease (KBILD) score and the University of California San Diego (UCSD) Shortness of Breath Questionnaire, and the presence and severity of small airway disease;
Variation of small airway dysfunction parameters in IPF patients after one year of antifibrotic treatment. | 1 year
  Evaluate presence and variation of small airway dysfunction parameters from the Single Breath Nitrogen (SBN2) test in IPF patients after one year of antifibrotic therapy.
Prevalence of tidal expiratory flow limitation at the time of diagnosis, before the initiation of antifibrotic therapy and after one year of antifibrotic treatment. | 1 year
  To evaluate the percentage of patients with IPF with tidal expiratory flow limitation measured by means of Negative Expiratory Pressure (NEP), at the time of diagnosis, before the initiation of antifibrotic therapy and after one year of therapy with antifibrotic treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Pulmonology Unit, ASST Santi Paolo e Carlo. Department of Health Sciences, University of Milan, Milan (Italy), Milan, Lombardy
  - Division of Respiratory Diseases, L. Sacco University Hospital, ASST Fatebenefratelli-Sacco, Milan, Italy. Department of Biomedical and Clinical Sciences, Università Degli Studi di Milano, Milano, Italy, Milan, Lombardy

IPD SHARING:
Plan to Share IPD: Undecided